CLINICAL TRIAL: NCT07329218
Title: Effect of Pelvic Floor Stretching on Pelvic Floor Myofascial Pain and Quality of Life in Postmenopausal Female
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AhmedAbdelhamid2025
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Floor Myofascial Pain
Keywords: postmenopausal female; pelvic floor myofascial pain; pelvic floor muscle stretching; pelvic floor muscle strengthening

STUDY DESIGN:
Intervention Model Description: Patients were randomized using the randomization block method into two groups, study (n=30) and control (n=30) groups. The allocation sequence was applied by a blinded and independent research assistant who opened sealed envelopes containing a computer-generated randomized number. study group received pelvic floor muscles stretching exercises while control group received Kegel exercises and pelvic rocking exercises.
Who Masked: Participant
Masking Description: Sixty female postmenopausal patients who had pelvic floor myofascial pain were chosen from the outpatient clinic of the Faculty of Physical Therapy, Delta University for Science and technology. education, occupation and duration of complaints of each patient. All were evaluated at the beginning of the treatment (week 0), at the endpoint of the treatment (week 4).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pelvic floor muscles Stretching (Experimental): The specification of the exercises are as follows Lie on the floor on the back. Slowly raise both the legs into the air. Hold the position for a few seconds. Slowly bring down the legs and then the knees as the patient return to the original resting position. Hold the position for 10 seconds and relax 30 seconds. Repeat 5 times. The exercises are performed for 10 minutes with warm up and cool down for duration of 10 minutes and for period of 4 weeks
  Interventions: Other: Pelvic floor muscles Stretching
- Kegel Exercise (Active Comparator): Patients will be in supine position with flexion of both lower limbs; they will be ordered to tighten perineum and anus for 10 seconds during inspiration, and then relaxed for 5~10 seconds during exhalation for ten times per session and this exercise will be repeated three times in a day
  Interventions: Other: Kegel Exercise
- Pelvic Rocking exercises (Active Comparator): The woman will be positioned on her hands and knees, with her hands placed directly under her shoulders and her knees under her hips. Then she will be asked to breathe in deeply, tuck her head downward, and round her back up, making a curve with her back in the shape of the letter C. Hold this position for a count of 6, then breathe out slowly and bring her head back up. Relax, keeping the back straight-don't allow it to curve toward the floor. Hold this for a count of 6, this exercise was done 8 times for min.
  Interventions: Other: Pelvic Rocking exercises

INTERVENTIONS:
Other: Kegel Exercise — already were described in arm descriptions
  Other Names: Pelvic floor muscles Stretching
  Arms: Kegel Exercise
Other: Pelvic Rocking exercises — already were described in arm descriptions
  Other Names: Pelvic floor muscles Stretching
  Arms: Pelvic Rocking exercises
Other: Pelvic floor muscles Stretching — already were described in arm descriptions
  Arms: Pelvic floor muscles Stretching

SUMMARY:
Menopause, also known as the climacteric, is the time when menstrual periods permanently stop, marking the end of reproduction, it typically occurs between the ages of 45 and 55, although the exact timing can vary, menopause is usually a natural change related to a decrease in circulating blood estrogen levels [1]. In the years before menopause, a woman's periods typically become irregular, which means that periods may be longer or shorter in duration or be lighter or heavier in the amount of flow. During this time, women often experience hot flashes; these typically last from 30 seconds to ten minutes and may be associated with shivering, night sweats, and reddening of the skin, while other symptoms may include vaginal dryness, trouble sleeping, and mood changes, the severity of symptoms varies between women [2].

Female pelvic floor muscles form a diaphragm that spans the entire pelvic cavity. They consist of the fibers of the coccygeus and the levator ani muscles, together with their fascia, the pelvic floor muscles provide support for the urethra, the vagina, and the rectum and constrict the urethral, vaginal, and anal orifices. Alterations in the composition of the pelvic floor muscles at menopause appear to affect their properties and, thereby, their ability to function adequately. This can lead to an increased prevalence in urinary incontinence and other lower urinary tract dysfunction, pelvic organ prolapses, and genitourinary syndrome of menopause [3].

During the menopausal transition, there is a substantial decrease in the number of ovarian follicles and numerous hormonal changes are observed. The first endocrine signal of the menopausal transition is a significant increase in follicle-stimulating hormone (FSH) levels. An important increase in FSH levels and a considerable decrease in estrogen and inhibin A concentrations are observed in the late stage of the menopausal transition. However, a 50% increase in FSH levels and a 50% decrease in estrogen concentrations are observed in the final postmenopausal period, these hormonal changes can directly affect pelvic floor muscle mass. After menopause, cross sectional areas of muscle mass decrease by 0.6% every year. Noncontractile muscle tissue mass (intramuscular fat mass) in postmenopausal women is two times greater that than in young women. The ratio of connective tissues to muscle fibrils in the urethral stricture and pelvic floor muscles decreases with age [4].

Non-surgical treatment of pelvic floor dysfunction mainly consists of manual approach, stimulation or relaxation techniques. Trigger points can be treated with local massage and stretching of the PFM. Using post isometric contraction techniques might help to give better stretching abilities of muscles [8]. In addition to manual manipulation, modalities such as electrostimulation, biofeedback, and vaginal dilators or vaginal weighted cones can be used to help with isolation of pelvic floor musculature and improve contraction. Electrical stimulation provides a small electrical current to contract the pelvic floor and assist the patient in isolation of the proper muscles. Biofeedback uses a vaginal or rectal pressure sensor to provide an audible and/or visual feedback of the strength of the muscle contraction. A vaginal weighted cone is inserted into the vagina and held in place by pelvic muscle contractions during activity Subjects and methods This study was a randomized controlled study. All procedures used in the study were compliant with the Declaration of Helsinki, which regulates research involving human subjects. Registration Clinical Trial Registration database (?) and approval from the Faculty of Physical Therapy, Delta University's institutional review board (F.P.T 250740). This study was carried out at an outpatient clinic at the Faculty of Physical Therapy, Delta University for Science and Technology, Egypt. The registration and recruitment of individuals and follow-up procedures were done from January 2025 to April 2025.

Subjects:

The patients were included in this study had these criteria: Females diagnosed with postmenopausal chronic pelvic pain between age group 45-55 years.

DETAILED DESCRIPTION:
Effect of pelvic floor stretching on pelvic floor myofascial pain and quality of life in postmenopausal female Menopause, also known as the climacteric, is the time when menstrual periods permanently stop, marking the end of reproduction, it typically occurs between the ages of 45 and 55, although the exact timing can vary, menopause is usually a natural change related to a decrease in circulating blood estrogen levels [1]. In the years before menopause, a woman's periods typically become irregular, which means that periods may be longer or shorter in duration or be lighter or heavier in the amount of flow. During this time, women often experience hot flashes; these typically last from 30 seconds to ten minutes and may be associated with shivering, night sweats, and reddening of the skin, while other symptoms may include vaginal dryness, trouble sleeping, and mood changes, the severity of symptoms varies between women [2].

Female pelvic floor muscles form a diaphragm that spans the entire pelvic cavity. They consist of the fibers of the coccygeus and the levator ani muscles, together with their fascia, the pelvic floor muscles provide support for the urethra, the vagina, and the rectum and constrict the urethral, vaginal, and anal orifices. Alterations in the composition of the pelvic floor muscles at menopause appear to affect their properties and, thereby, their ability to function adequately. This can lead to an increased prevalence in urinary incontinence and other lower urinary tract dysfunction, pelvic organ prolapses, and genitourinary syndrome of menopause [3].

During the menopausal transition, there is a substantial decrease in the number of ovarian follicles and numerous hormonal changes are observed. The first endocrine signal of the menopausal transition is a significant increase in follicle-stimulating hormone (FSH) levels. An important increase in FSH levels and a considerable decrease in estrogen and inhibin A concentrations are observed in the late stage of the menopausal transition. However, a 50% increase in FSH levels and a 50% decrease in estrogen concentrations are observed in the final postmenopausal period, these hormonal changes can directly affect pelvic floor muscle mass. After menopause, cross sectional areas of muscle mass decrease by 0.6% every year. Noncontractile muscle tissue mass (intramuscular fat mass) in postmenopausal women is two times greater that than in young women. The ratio of connective tissues to muscle fibrils in the urethral stricture and pelvic floor muscles decreases with age [4].

Myofascial pelvic pain described as myalgia condition with local and referred pain patterns, it refers to pain found in the pelvic floor musculature and the connecting fascia. It is characterized by adverse symptoms of tender points, myofascial trigger points in skeletal muscles [5].

Pelvic floor myofascial pain was common in patients seeking evaluation for pelvic floor disorder symptoms. Location and severity of pelvic floor myofascial pain was significantly correlated with degree of symptom bother, even after controlling for postmenopausal status. Given the high prevalence of pelvic floor myofascial pain in these patients and correlation between pain severity and degree of symptom bother, a routine assessment for pelvic floor myofascial pain should be considered for all patients presenting for evaluation of pelvic floor symptoms [6].

The World Health Organization (WHO) defines QoL as "an individual's perception of their position in life, in the context of the culture and value system in which they live, and in relation to their goals, expectations, standards, and concerns". Fifty to 80% of women complain about menopausal symptoms such as hot flashes, night sweats, sleep disturbances, tiredness, and depression, they are the principal determinants of a reduced health-related quality of life (HRQL), which is detectable soon after the onset of menopause, menopause-related symptoms have a negative impact on the QoL of perimenopausal women. Budakoglu et al, showed that the QoL in postmenopausal women is worse than that of premenopausal women [7].

Non-surgical treatment of pelvic floor dysfunction mainly consists of manual approach, stimulation or relaxation techniques. Trigger points can be treated with local massage and stretching of the PFM. Using post isometric contraction techniques might help to give better stretching abilities of muscles [8]. In addition to manual manipulation, modalities such as electrostimulation, biofeedback, and vaginal dilators or vaginal weighted cones can be used to help with isolation of pelvic floor musculature and improve contraction. Electrical stimulation provides a small electrical current to contract the pelvic floor and assist the patient in isolation of the proper muscles. Biofeedback uses a vaginal or rectal pressure sensor to provide an audible and/or visual feedback of the strength of the muscle contraction. A vaginal weighted cone is inserted into the vagina and held in place by pelvic muscle contractions during activity [9].

The pelvic floor can be made stronger by performing Kegel exercises, which involve regularly tightening and relaxing the muscles that make up the pelvic floor. Exercises designed by Kegel are regarded as a crucial part of pelvic floor muscle rehabilitation. Performing Kegel's exercise and stretching regularly helps enhance the function of the pelvic floor muscles. There was an effect of pelvic floor muscle exercise and stretching to reducing the pain and improving quality of life in young women with primary dysmenorrhea [10].

Pelvic floor muscle training (PFMT) refers to exercises for improving PFM strength, endurance, power and/or relaxation. It is taught and monitored by health professionals such as physiotherapists. PFMT was proven to be effective in the treatment of urinary incontinence and pelvic organ prolapses. With its low-cost and minimal adverse effects, it is recommended as first-line treatment for pelvic floor dysfunctions [11].

So, this study aims to investigate the difference between the effect of pelvic floor muscles strengthening exercise and stretching in reducing the pain and improving quality of life in postmenopausal women.

Subjects and methods This study was a randomized controlled study. All procedures used in the study were compliant with the Declaration of Helsinki, which regulates research involving human subjects. Registration Clinical Trial Registration database (?) and approval from the Faculty of Physical Therapy, Delta University's institutional review board (F.P.T 250740). This study was carried out at outpatient clinic at faculty of physical therapy, delta university for science and technology, Egypt. The registration and recruitment of individuals and follow-up procedures were done from January 2025 to April 2025.

Subjects:

The patients were included in this study had these criteria: Females diagnosed with postmenopausal chronic pelvic pain between age group 45-55 years.

The exclusion criteria: history of pelvic inflammatory disease, endometriosis, any pathology, compulsory use of special drugs, had symptoms such as (tingling, itching, discharge), use of painkillers during the study period, any musculoskeletal problems causing inability to perform pelvic floor strengthening or stretching exercises, mental, psychological problems.

Sample size A convenient sample of 70 participants were screened for study eligibility. The sample size was calculated utilizing G*Power based on a prior study with an effect size of 0.8. to detect a true difference in means with 80% power and a 5% significance level. An estimated sample size of 60 patients were randomly allocated to a software application. Group A (the study group) Kegel strengthening exercises and pelvic rocking exercise combined with pelvic stretching exercises for pelvic floor muscles. The 2nd group (group B, control group) received Kegel strengthening exercises and pelvic rocking exercise for pelvic floor muscles.

Randomization Informed consent was attained from each individual after explanation of the aim as well as benefits of the study. Individuals were informed about the privacy of their information and their right to stop or withdraw at any time. They were randomized using the randomization block method into two groups, study (n=30) and control (n=30) groups. Allocation sequence was applied by a blinded and independent research assistant who opened sealed envelopes containing a computer-generated randomized number.

Assessment procedures:

The assessors who participated in this study were blinded to the patients' allocation in the studied groups. The outcome measures of this study were evaluated by one physiotherapist with an experience of more than 20 years in musculoskeletal and neurological conditions. Evaluating the pain severity and quality of life measures were conducted for all patients before commencing the treatment and immediately after completing the treatment period of 4 weeks in the following order:

1. Pain severity for pelvic floor myofascial pain:

   We used Visual Analogue Scale (VAS) which is a reliable and effective tool of pain intensity that is sensitive to variations in pain caused by clinical conditions, was used to assess the severity of the pain. At the scale's left end, a zero means there is no pain, and a 10 means the most agonizing suffering possible. A minor improvement with a change of 1.1-1.2 cm is clinically meaningful [12].
2. Quality of life assessment:

We used The Menopause Specific Quality of Life Questionnaire (MENQOL):

It was developed by (Hilditch et al., 1996). using a sample of women 47-62 years old who had ceased menstruation for 2-7 years, who had not had a hysterectomy, and who had not used hormone therapy during the preceding 6 months. It is a validated questionnaire for the assessment of menopausal women's symptoms and an effective instrument. The questionnaire consists of 29 sub-items with a 7-point scale from 0 to 6, and includes four domains: vasomotor, psychosocial, physical, and sexual [13].

Intervention procedures:

Kegel Exercise Patients will be in supine position with flexion of both lower limbs, they will be ordered to tighten perineum and anus for 10 seconds during inspiration, and then relaxed for 5~10 seconds during exhalation for ten times per session and this exercise will be repeated three times in a day [14].

Pelvic Rocking: This exercise strengthens the back, hip, and abdominal muscles. The woman will be positioned on her hands and knees, with her hands will be placed directly under her shoulders and the knees under the hips. Then she will be asked to breathe in deeply, tuck her head downward and round her back up, making a curve with her back in the shape of the letter C. Hold this position for a count of 6, then breathe out slowly and bring her head back up. Relax, keeping the back straight-don't allow it to curve toward the floor. Hold this for a count of 6, this exercise was done 8 times for 5min. [15].

Pelvic Stretching: The specification of the exercises are as follows Lie on the floor on the back. Slowly raise both the legs into the air. Hold the position for a few seconds. Slowly bring down the legs and then the knees as the patient return to the original resting position. Hold the position for 10 seconds and relax 30 seconds. Repeat 5 times. The exercises are performed for 10 minutes with warm up and cool down for duration of 10 minutes and for period of 4 weeks [1].

ELIGIBILITY:
Inclusion Criteria:

* Females diagnosed with postmenopausal chronic pelvic pain between the ages of 45 and 55 years

Exclusion Criteria: history of pelvic inflammatory disease, endometriosis, any pathology, compulsory use of special drugs, having symptoms such as tingling, itching, or discharge, use of painkillers during the study period, any musculoskeletal problems causing inability to perform pelvic floor strengthening or stretching exercises, mental, psychological problems.

-

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — our study on postmenopausal females so it is gender based
Enrollment: 60 (Actual)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
1- Pain severity for pelvic floor myofascial pain | pre the intervention and immediately after the intervention
  Visual Analogue Scale (VAS) which is a reliable and effective tool of pain intensity that is sensitive to variations in pain caused by clinical conditions, was used to assess the severity of the pain. At the scale's left end, a zero means there is no pain, and a 10 means the most agonizing suffering possible. A minor improvement with a change of 1.1-1.2 cm is clinically meaningful
Quality of life assessment | pre the intervention and immediately after the intervention
  The Menopause Specific Quality of Life Questionnaire (MENQOL):
  It was developed by (Hilditch et al., 1996). using a sample of women 47-62 years old who had ceased menstruation for 2-7 years, who had not had a hysterectomy, and who had not used hormone therapy during the preceding 6 months. It is a validated questionnaire for the assessment of menopausal women's symptoms and an effective instrument. The questionnaire consists of 29 sub-items with a 7-point scale from 0 to 6, and includes four domains: vasomotor, psychosocial, physical, and sexual

CONTACTS AND LOCATIONS:
Locations (1):
- Horus University, Damietta, Egypt